CLINICAL TRIAL: NCT03385005
Title: Evaluating Neuromuscular Stimulation for Restoring Hand Movements
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Chad Bouton, Vice President, Advanced Engineering; Bioelectronic Medicine, Northwell Health
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: 17-0070
Record Dates: First submitted 2017-09-26; First posted 2017-12-28 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers; Spinal Cord Injury Cervical; Physical and Rehabilitation Medicine
Keywords: Physical and Rehabilitation Medicine; Transcutaneous Electrical Nerve Stimulation; Healthy Volunteer; Spinal Cord Injury; Biomedical Engineering
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: The study will involve 3-10 eligible healthy volunteers and 2-5 eligible individuals with a stable cervical spinal cord injury. The study will first enroll healthy volunteers into the study in order to determine the feasibility of evoking refined hand movements through electrical stimulation, and determine the electrical stimulation parameters and electrode spatial configurations responsible for various hand movements. After this is done, the study will proceed with the enrollment of individuals with spinal cord injuries. This enrollment process is being done to reduce the participation time required for participants with a spinal cord injury, and thus lower the likelihood of risks that are more prevalent among individuals with a spinal cord injury.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Healthy Volunteers (Active Comparator): This arm consists of healthy volunteers receiving electrical stimulation of the muscles within the forearm via an investigational (not FDA approved) neuromuscular stimulator.
  Interventions: Device: Participants will receive neuromuscular electrical stimulation via an investigational (not FDA approved) neuromuscular stimulator.
- Spinal Cord Injury Participants (Active Comparator): This arm consists of spinal cord injury participants receiving electrical stimulation of the muscles within the forearm via an investigational (not FDA approved) neuromuscular stimulator.
  Interventions: Device: Participants will receive neuromuscular electrical stimulation via an investigational (not FDA approved) neuromuscular stimulator.

INTERVENTIONS:
Device: Participants will receive neuromuscular electrical stimulation via an investigational (not FDA approved) neuromuscular stimulator. — The study involves the administration of various electrical pulses being delivered to muscles of the forearm from a neuromuscular stimulator in order to evoke different hand and finger movements. The grip strength and evoked forces at the fingertips will also be measured using sensors.

SUMMARY:
The specific aim of this study is to evoke functional movement in the hand of both healthy individuals and individuals diagnosed with a stable cervical spinal cord injury with non-functional movement of the fingers. The primary purpose of this study is to determine the feasibility of achieving refined hand movements through electrical stimulation of the muscles within the forearm. It is believed that this study will be able to identify specific stimulation parameters and electrode spatial configurations responsible for various refined hand movements.

After an eligible individual agrees to participate in this study, s/he will receive transcutaneous electrical stimulation on the forearm in order to evoke different hand and finger movements. The precision, specificity, and extent of these movements will be visually assessed. In order to better evaluate these movements, participants may also be asked to perform various functional tasks with their hand. The grip strength and evoked forces at the fingertips will also be measured using sensors. There will be up to 4 study sessions each week for up to 8 weeks, with each session lasting up to 4 hours. Upon completion of these study sessions, the individual's participation in the study is considered complete.

DETAILED DESCRIPTION:
In order to evaluate whether electrical stimulation applied to the muscles within the forearm can evoke functional movement in the hand, participants will receive transcutaneous electrical stimulation via an investigational (not FDA approved) neuromuscular stimulator.

Participants will be asked to attend up to 4 study sessions a week for up to 8 weeks, with each session lasting up to 4 hours. At these sessions, electrical pulses will be sent to the forearm muscles through electrodes placed on the skin. These electrodes may also be accompanied with a gel or lotion to allow for a better connection of the electrodes to the skin. The precision, specificity, and extent of hand and finger movements will be visually assessed in real time and later reassessed on video recordings of the session. The study will also involve the placement of sensors on the hand and finger to measure the amount of grip strength and evoked forces. In order to monitor the health of participants, the study will assess blood pressure and heart rate before, during, and after the electrical stimulation. Upon completion of these study sessions, the individual's participation in the study is considered complete.

ELIGIBILITY:
Inclusion Criteria for Health Volunteers:

* Individuals between 18 and 65 years of age
* Individuals without physical disabilities or conditions/diseases that may make them incapable of completing the physical study tasks or otherwise places them at a greater risk of harm
* Individuals that are considered English Proficient due to the study requirements to follow verbal commands during testing sessions
* Individuals that are able to comprehend the study goals and procedures, and are able to provide informed consent for participation
* Individuals that are willing and able to visit the study center for study procedures, which will be up to 4 sessions a week for up to 8 weeks at up to 4 hours per session
* Have the ability and willingness to undergo upper limb electrodiagnostic and nerve conduction studies
* Demonstrate typical amplitude, latency, and conduction velocity in the distal median, ulnar, and radial nerves of at least one upper limb

Exclusion Criteria for Healthy Volunteers:

* Individuals participating in another research study that may affect the conduct or results of this study
* Individuals having or exhibiting any of the following:

  * Stage III-IV pressure ulcers
  * Chronically-implanted electronic medical device (e.g. baclofen pump, deep brain stimulator, epidural stimulator, cardiac pacemaker, vagus nerve stimulator, or other)
  * Prior tendon transfer to enhance hand function
  * History of autoimmune disease
  * Cancer
  * Biochemical abnormalities of the liver, kidney, or pancreas
  * Prior difficulties or allergy to general anesthesia
  * Ventilator dependence
  * History of serious mood or thought disorder
  * Significant residual clinically evident traumatic brain injury or cognitive impairment
  * Uncontrolled autonomic dysreflexia
  * Spasticity in the upper extremities that is uncontrolled by pharmacological methods
* Individuals with a substance abuse (alcoholism or other) problem
* Pregnant women
* Prisoners

Inclusion Criteria for Participants with a Spinal Cord Injury:

* Individuals between 18 and 65 years of age
* Individuals with a stable cervical spinal cord injury with ISNCSCI motor scores for fingers of 0 - 2 (non-functional), and at least one year from initial spinal cord injury
* Individuals that are considered English Proficient due to the study requirements to follow verbal commands during testing sessions
* Individuals that are able to comprehend the study goals and procedures, and are able to provide informed consent for participation
* Individuals that are willing and able to visit the study center for study procedures, which will be up to 4 sessions a week for up to 8 weeks at up to 4 hours per session
* Have the ability and willingness to undergo upper limb electrodiagnostic and nerve conduction studies
* Demonstrate typical amplitude, latency, and conduction velocity in the distal median, ulnar, and radial nerves of at least one upper limb (as expected for a person at their stage of time post spinal cord injury)

Exclusion Criteria for Participants with a Spinal Cord Injury:

* Individuals participating in another research study that may affect the conduct or results of this study
* Individuals having or exhibiting any of the following:

  * Stage III-IV pressure ulcers
  * Chronically-implanted electronic medical device (e.g. baclofen pump, deep brain stimulator, epidural stimulator, cardiac pacemaker, vagus nerve stimulator, or other)
  * Prior tendon transfer to enhance hand function
  * History of autoimmune disease
  * Cancer
  * Biochemical abnormalities of the liver, kidney, or pancreas
  * Prior difficulties or allergy to general anesthesia
  * Ventilator dependence
  * History of serious mood or thought disorder
  * Significant residual clinically evident traumatic brain injury or cognitive impairment
  * Uncontrolled autonomic dysreflexia
  * Spasticity in the upper extremities that is uncontrolled by pharmacological methods
* Individuals with a substance abuse (alcoholism or other) problem
* Pregnant women
* Prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study is to determine the feasibility of achieving refined hand movements through electrical stimulation of the muscles within the forearm, as assessed by visual inspection. | This outcome measure will be assessed at each study session throughout the 8-week duration of the study.
  The primary outcome measure will be achievable wrist and finger movements that will be visually assessed for the type and extent of motion in relation to the stimulation parameters and electrode spatial configurations. The extent of wrist, forearm, and individual finger movements will be categorized as either flexion, extension, adduction, abduction, pronation, or supination and graded as no movement, slight movement, moderate movement, or substantial movement.
The primary outcome of the study is to determine the feasibility of achieving refined hand movements through electrical stimulation of the muscles within the forearm, as assessed by force sensors. | This outcome measure will be assessed at each study session throughout the 8-week duration of the study.
  The primary outcome measure will be achievable wrist and finger movements that will be assessed by the exerted force (measured in Newtons by force sensors on the fingers and palm) in each of the flexion, extension, adduction, abduction, pronation, or supination movements. This will provide the magnitude of the movement in relation to the stimulation parameters and electrode spatial configurations.

CONTACTS AND LOCATIONS:
Overall Officials: Chad E Bouton, MS, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health's The Feinstein Institute for Medical Research, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The identifiable information collected on this study will only be shared with other researchers that have obtained approval from the institutional review board (IRB). After a request for study information is received, the principal investigator (Chad Bouton, MS) will determine whether the requested information can be shared given the authorization status of the study participants. After approval by the principal investigator, the researcher will be required to present a letter indicating IRB approval of their study and a copy of the approved protocol indicating that approval includes the receipt of information from this study. If this information is obtained, the principal investigator will provide the requested information (taking into account the authorization status of participants) to the researchers in a HIPAA-compliant manner.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study will only provide identifiable information pertaining to participants as long as there is active and valid IRB approval of the study. After the study is completed and the study has been closed with the IRB, information will no longer be shared.
Access Criteria: The study will only share information with other researchers that have been approved by the principal investigator (Chad Bouton, MS), have showed evidence that their study has valid IRB approval that includes the ability to receive the requested information, and has provided a copy of the approved protocol to verify they can receive the requested information and that the information will be stored in a HIPAA-compliant manner.

REFERENCES:
- [Background] Bouton CE, Shaikhouni A, Annetta NV, Bockbrader MA, Friedenberg DA, Nielson DM, Sharma G, Sederberg PB, Glenn BC, Mysiw WJ, Morgan AG, Deogaonkar M, Rezai AR. Restoring cortical control of functional movement in a human with quadriplegia. Nature. 2016 May 12;533(7602):247-50. doi: 10.1038/nature17435. Epub 2016 Apr 13. PMID 27074513
- [Derived] Bhagat N, King K, Ramdeo R, Stein A, Bouton C. Determining grasp selection from arm trajectories via deep learning to enable functional hand movement in tetraplegia. Bioelectron Med. 2020 Aug 25;6:17. doi: 10.1186/s42234-020-00053-5. eCollection 2020. PMID 32864392
- [Derived] Ciancibello J, King K, Meghrazi MA, Padmanaban S, Levy T, Ramdeo R, Straka M, Bouton C. Closed-loop neuromuscular electrical stimulation using feedforward-feedback control and textile electrodes to regulate grasp force in quadriplegia. Bioelectron Med. 2019 Nov 1;5:19. doi: 10.1186/s42234-019-0034-y. eCollection 2019. PMID 32232108
- See also: Restoring Cortical Control of Functional Movement in a Human with Quadriplegia — https://www.nature.com/nature/journal/v533/n7602/full/nature17435.html